CLINICAL TRIAL: NCT06652555
Title: The CNS AE of Lorlatinib in Patients with ALK-positive Advanced NSCLC
Brief Title: The Incidence and Risk Factors of Central Nervous System Adverse Events of Lorlatinib in Patients with ALK-positive Advanced Non-small Cell Lung Cancer: a Real-world Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chunxia Su, Director of Clinical Research Center, Shanghai Pulmonary Hospital, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2024LY0856
Record Dates: First submitted 2024-09-29; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: ALK; NSCLC
Keywords: ALK; NSCLC

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group 1: Baseline characteristics and information during loratinib treatment were collected
  Interventions: Other: Group 1

INTERVENTIONS:
Other: Group 1 — without Intervention

SUMMARY:
The goal of this study is to investigate the incidence and risk factors of central nervous system adverse events of Lorlatinib in patients with ALK-positive advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
The goal of this study is to investigate the incidence and risk factors of central nervous system adverse events of Lorlatinib in patients with ALK-positive advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced (stage IIIb/IIIc), metastatic, or recurrent (stage IV) NSCLC confirmed by histology or cytology, who are not eligible for curative surgery and cannot undergo definitive radiotherapy/chemotherapy, according to the 8th edition of the TNM staging classification by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer;
* ALK-positive and the test results were based on RT-PCR /FISH /IHC /NGS methods in the laboratory department or testing institution of the hospital
* receiving targeted therapy with Lorlatinib
* age ≥18 years old
* follow-up after receipt of Lorlatinib
* voluntarily participate in the study and sign informed consent

Exclusion Criteria:

* evidence of any severe or uncontrolled systemic illness, including uncontrolled hypertension and active bleeding, active infections including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
* combined with other malignant tumors and received other anti-tumor therapy during the treatment of Lorlatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK-positive NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2026-09-29 (Estimated); Study Completion 2027-09-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of central nervous system (CNS) adverse events (AEs) associated with lorlatinib in real world study. | 2 year
  The incidence of central nervous system (CNS) adverse events (AEs) associated with lorlatinib will be reported, such as cognitive effects, mood effects, speech effects and psychotic effects.

SECONDARY OUTCOMES:
To explore the optimized therapy management strategies for CNS AEs associated with lorlatinib in real-world study. | 1 year
  According to the data from CROWN study, management strategies such as to dose interruption, dose reduction or concurrent medication would minimize the impact of CNS AEs effects. However, the optimized therapy management strategies for CNS AEs associated with lorlatinib in real-world study of China needs to be further clarified.
Analysis of factors associated with developing CNS AEs related to lorlatinib treatment. | 1 year
  The association between baseline characteristics and CNS adverse effects will be evaluated. Baseline characteristics include age, gender, medical history, brain metastases at baseline, previous brain radiation, and lorlatinib treatment lines, among others.
Correlation analysis between CNS AEs occurrence and anti-tumor efficacy | 24 weeks
  Landmark analysis will be used to investigate the possible association between development of CNS AEs within 24 weeks of initiating lorlatinib and progression-free survival (PFS) as well as the objective response rate (ORR).

CONTACTS AND LOCATIONS:
Overall Officials: Chunxia Su, Doctor, Study Chair — Shanghai Pulmonary Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
research article
Supporting Information: Study Protocol
Time Frame: up to 36 month
Access Criteria: Send an email requesting research